CLINICAL TRIAL: NCT01680094
Title: The Safety and Efficacy of The Histone Deacetylase Inhibitor Panobinostat for Purging HIV-1 From The Latent Reservoir (CLEAR) Study
Brief Title: Safety and Effect of The HDAC Inhibitor Panobinostat on HIV-1 Expression in Patients on Suppressive HAART
Acronym: CLEAR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Massachusetts General Hospital (Other); Monash University (Other); University of Sydney (Other); Novartis (Industry); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEAR0001
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: HIV Infection
Keywords: HIV Infection; Panobinostat; Lentivirus Infections; Retroviridae Infections; RNA Virus Infections; Virus Diseases; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases; Immunologic Deficiency Syndromes; Immune System Diseases; Histone Deacetylase Inhibitors; Therapeutic Uses
MeSH Terms: conditions — HIV Infections; Lentivirus Infections; Retroviridae Infections; RNA Virus Infections; Virus Diseases; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases; Immunologic Deficiency Syndromes; Immune System Diseases | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Panobinostat (Experimental): 20 mg panobinostat will be administered orally on days 1, 3, and 5 (TIW) every other week (QOW) for a period of 8 weeks while maintaining background HAART
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat — 20 mg panobinostat will be administered orally on days 1, 3, and 5 (TIW) every other week (QOW) for a period of 8 weeks while maintaining background HAART
  Other Names: LBH589

SUMMARY:
The purpose of this study is to assess the safety and ability of panobinostat to re-activate HIV transcription in latently infected CD4+ T-cells among HIV-infected patients on stable antiretroviral therapy

DETAILED DESCRIPTION:
Despite effective highly active antiretroviral treatment (HAART), HIV-infection persists and rebounds upon treatment interruption, presumably due to latently infected resting CD4+ T-cells. To achieve eradication of HIV-infection this reservoir of latently HIV-infected cells must be depleted.

Several therapeutic strategies are considered in HIV-cure related research. One approach is to exploit the ability of histone deacetylase (HDAC) inhibitors to reactivate HIV-1 expression in latently infected cells in the presence of HAART.

This is an investigator initiated single-group, non-randomized interventional phase I/II trial designed to evaluate the safety and ability of oral panobinostat to activate HIV-transcription in latently infected CD4+ T-cells of HIV-infected patients on suppressive HAART. The study will enrol 16 patients. Each subject will be used as his/her own control in a before-after design: endpoints measured after study intervention will be compared to baseline for each subject.

The main study will comprise three phases:

1. A pre-treatment screening/observation phase of 4 weeks (weeks 0-4)
2. A treatment phase of 8 weeks (weeks 4-12), where 20 mg panobinostat will be administered orally on days 1, 3, and 5 (TIW) every other week (QOW) while maintaining background HAART (co-therapy)
3. A post-treatment follow-up phase of 24 weeks (weeks 12-36) to evaluate the effect of study treatment

Study participants will be reviewed 13 times during the course of study treatment and follow-up. Blood will be drawn for HIV viral load assessments, CD4 cell counts, biochemistry, hematology and additional immunological and virological analyses. An electrocardiogram of the heart (ECG) will be taken at screening, day 10 and 24 post treatment initiation.

The safety and tolerability of panobinostat will be evaluated based on physical exams, laboratory tests and questions about any problems patients may have experienced during the study. A pre-specified schedule based will guide dose modification in case of unacceptable adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Age >18 years
* HIV-1 plasma RNA <50 copies/ml for at least 2 years with at least 2 viral load measures per year. Episodes of a single HIV plasma RNA 50-199 copies/ml will not exclude participation if the subsequent HIV plasma RNA was <50 copies/ml
* Receiving HAART, defined as at least 2 nucleoside/nucleotide reverse transcriptase inhibitors plus a non-nucleoside reverse transcriptase inhibitor, integrase inhibitor, or a protease inhibitor
* CD4+ T-cell count >500/mm3 on minimum 2 occasions in the last 12 months prior to study entry
* Able to give informed consent

Exclusion Criteria:

* Any significant acute medical illness in the past 8 weeks
* Any evidence of an active AIDS-defining opportunistic infection
* Current or recent gastrointestinal disease that may impact the absorption of the investigational drug
* Any gastrointestinal surgery that could impact upon the absorption of the investigational drug
* Active alcohol or substance use that, in the Investigator's opinion, will prevent adequate compliance with study therapy
* Patient has the following laboratory values within 3 weeks before starting the investigational drug (lab tests may be repeated, as clinically indicated, to obtain acceptable values before failure at screening is concluded but supportive therapies are not to be administered within the week prior to screening tests for ANC or platelet count)

  * Hepatic transaminases (AST or ALT) ≥3 x upper limit of normal (ULN)
  * Serum total bilirubin ≥1.5 ULN
  * Serum creatinine levels ≥1.5 x ULN, or calculated creatinine clearance ≤60 ml/min
  * Platelet count ≤100 x109/L
  * Absolute neutrophil count ≤1.5x109/L
  * Serum potassium, magnesium, phosphorus outside normal limits
  * Total calcium (corrected for serum albumin) or ionized calcium ≤lower normal limits
* Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood
* A personal history of clinically significant cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for Torsades de pointes (e.g. heart failure)
* History of malignancy or transplantation, including skin cancers or Kaposi sarcoma
* History of diabetes mellitus
* Use of a protease inhibitor
* Receipt of immunomodulating agents, immunization or systemic chemotherapeutic agents within 28 days prior to study entry
* Use of an agent definitely or possibly associated with effects on QT intervals within 2 weeks of screening
* ECG at screening that shows QTc >450 msec when calculated using the Fridericia formula from either lead V3 or V4
* Known resistance to >2 classes of ART
* Known hypersensitivity to the components of panobinostat or its analogues
* Current use of sodium valproate or other HDAC inhibitor
* Women who are pregnant or breastfeeding, or with a positive pregnancy test during screening or Women of Child Bearing Potential (WOCBP) who are unwilling or unable to use an acceptable method of contraception (according to the Danish Medicines Agency guidelines) to avoid pregnancy for the entire study period and for at least 4 weeks before and 4 weeks after study treatment
* Males or females who are unwilling or unable to use barrier contraception during sexual intercourse for the entire study period, including at least 4 weeks before, 4 weeks after study treatment, and when plasma HIV-RNA is detectable using standard assays

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HIV transcription in latently infected CD4+ T-cells as measured by copies of unspliced HIV-RNA in the CD4+ T-cells of HIV-infected patients on suppressive HAART | Day 1 (before study drug and 2 hours after first dose), Day 2, 5, 10, 15, 24, 29, 38, 43, 52

SECONDARY OUTCOMES:
Change from baseline in the size of the latent HIV-reservoir as measured by copies of proviral HIV-DNA per 10⁶ CD4+ T-cells | 12 and 32 weeks after initiation of study treatment
Change from baseline in the frequency of cells latently infected with replication competent HIV expressed as infectious units per million (IUPM) | 12 weeks after initiation of study treatment
Safety evaluation, as measured by adverse events (AE), adverse reactions (AR), serious adverse events (SAE), serious adverse reactions (SAR), and serious unexpected serious adverse reactions (SUSAR) | Active follow-up until 32 weeks after initiation of study treatment
Plasma HIV-RNA as measured by the single copy assay | Day 1 (before study drug and 2 hours after first dose), Day 2, 5, 10, 15, 24, 29, 38, 43, 52, 84, 224
During an optional HAART-interruption study (if performed, see below): 1) Time to viremia >1000 copies/ml; 2) Time to meet criteria to restart HAART | To be performed upon completion of 32 weeks follow-up based on the below specified criteria
  Upon completion of the study, subjects may be invited to participate in an additional observational study in which HAART will be interrupted to evaluate the effect of study treatment on virological control. Enrolment into this study is optional and conditioned by the following criteria pertaining to the effect of study treatment on the latent HIV-1 reservoir:
  * Significant increase in unspliced HIV-RNA during in accordance with the primary endpoint measure
  * CD4+ T-cell count >500/mm3

CONTACTS AND LOCATIONS:
Overall Officials: Lars Østergaard, MD,DMSc,PhD, Study Director — Aarhus University Hospital; Thomas A Rasmussen, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Infectious Diseases, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Corley MJ, Pang APS, Rasmussen TA, Tolstrup M, Sogaard OS, Ndhlovu LC. Candidate host epigenetic marks predictive for HIV reservoir size, responsiveness to latency reversal, and viral rebound. AIDS. 2021 Nov 15;35(14):2269-2279. doi: 10.1097/QAD.0000000000003065. PMID 34482353
- [Derived] Garrido C, Tolstrup M, Sogaard OS, Rasmussen TA, Allard B, Soriano-Sarabia N, Archin NM, Margolis DM. In-vivo administration of histone deacetylase inhibitors does not impair natural killer cell function in HIV+ individuals. AIDS. 2019 Mar 15;33(4):605-613. doi: 10.1097/QAD.0000000000002112. PMID 30830886
- [Derived] Bjerg Christensen A, Dige A, Vad-Nielsen J, Brinkmann CR, Bendix M, Ostergaard L, Tolstrup M, Sogaard OS, Rasmussen TA, Randel Nyengaard J, Agnholt J, Denton PW. Administration of Panobinostat Is Associated with Increased IL-17A mRNA in the Intestinal Epithelium of HIV-1 Patients. Mediators Inflamm. 2015;2015:120605. doi: 10.1155/2015/120605. Epub 2015 Dec 1. PMID 26696749
- [Derived] Rasmussen TA, Tolstrup M, Brinkmann CR, Olesen R, Erikstrup C, Solomon A, Winckelmann A, Palmer S, Dinarello C, Buzon M, Lichterfeld M, Lewin SR, Ostergaard L, Sogaard OS. Panobinostat, a histone deacetylase inhibitor, for latent-virus reactivation in HIV-infected patients on suppressive antiretroviral therapy: a phase 1/2, single group, clinical trial. Lancet HIV. 2014 Oct;1(1):e13-21. doi: 10.1016/S2352-3018(14)70014-1. Epub 2014 Sep 15. PMID 26423811